CLINICAL TRIAL: NCT03726307
Title: Allogeneic Regulatory Dendritic Cell (DCreg) Therapy in Live-Donor Renal Transplant Recipients
Brief Title: Allogeneic Regulatory Dendritic Cell (DCreg) Renal Study
Acronym: RTB-006
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Angus W. Thomson PhD DSc (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Angus W. Thomson PhD DSc, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19040393; U01AI136779 (NIH)
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplant; Renal Transplant Recipients
Keywords: donor recipient pairs; allogeneic regulatory dendritic cell therapy (DCreg); DCreg therapy; de novo (first) live-donor renal transplant recipients

STUDY DESIGN:
Intervention Model Description: Open-label, dose-escalation, phase 1 clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- DCreg: 0.5 million cells/kg+SOC (Experimental): N=3 participants will receive 0.5 (± 0.1) million cells/kg body weight as a single infusion.
  Standard of Care (SOC) immunosuppressive agents (ISA): Participants will receive combination ISA according to the site's SOC regimen, with two exceptions:
  * mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
  * the pre-transplant dose of MPA will be half the standard post-transplant dose due to increased drug bioavailability in recipients with low glomerular filtration rate (GFR).
  Participants will be maintained on triple IS therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.
  Interventions: Biological: DCreg: 0.5 million cells/kg+SOC
- DCreg: 1.2 million cells/kg+SOC (Experimental): N=3 participants will receive 1.2 (± 0.2) million cells/kg body weight as a single infusion.
  Standard of Care (SOC) immunosuppressive agents (ISA): Participants will receive combination ISA according to the site's SOC regimen, with two exceptions:
  * mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
  * the pre-transplant dose of MPA will be half the standard post-transplant dose due to increased drug bioavailability in recipients with low glomerular filtration rate (GFR).
  Participants will be maintained on triple IS therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.
  Interventions: Biological: DCreg: 1.2 million cells/kg+SOC
- DCreg:2.5 to 5.0 million cells/kg+SOC (Experimental): N=8 participants will receive 25 to 5.0 million cells /kg body weight as a single infusion.
  Standard of Care (SOC) immunosuppressive agents (ISA): Participants will receive combination ISA according to the site's SOC regimen, with two exceptions:
  * mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
  * the pre-transplant dose of MPA will be half the standard post-transplant dose due to increased drug bioavailability in recipients with low glomerular filtration rate (GFR).
  Participants will be maintained on triple IS therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.
  Interventions: Biological: DCreg:2.5 to 5.0 million cells/kg+SOC

INTERVENTIONS:
Biological: DCreg: 0.5 million cells/kg+SOC — DCreg 0.5 (±0.1) million cells/kilogram body weight infused as a single dose.
  Standard of Care (SOC) immunosuppressive agents (ISA): Participants will receive combination ISA according to the site's SOC regimen, with two exceptions:
  * mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
  * the pre-transplant dose of MPA will be half the standard post-transplant dose due to increased drug bioavailability in recipients with low glomerular filtration rate (GFR).
  Participants will be maintained on triple IS therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.
  Other Names: Regulatory Donor-Derived Dendritic Cells (DCreg)
  Arms: DCreg: 0.5 million cells/kg+SOC
Biological: DCreg: 1.2 million cells/kg+SOC — DCreg 1.2 (±02) million cells/kilogram body weight infused as a single dose.
  Standard of Care (SOC) immunosuppressive agents (ISA): Participants will receive combination ISA according to the site's SOC regimen, with two exceptions:
  * mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
  * the pre-transplant dose of MPA will be half the standard post-transplant dose due to increased drug bioavailability in recipients with low glomerular filtration rate (GFR).
  Participants will be maintained on triple IS therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.
  Other Names: Regulatory Donor-Derived Dendritic Cells (DCreg)
  Arms: DCreg: 1.2 million cells/kg+SOC
Biological: DCreg:2.5 to 5.0 million cells/kg+SOC — DCreg 2.5 to 5.0 million cells/kilogram body weight infused as a single dose.
  Standard of Care (SOC) immunosuppressive agents (ISA): Participants will receive combination ISA according to the site's SOC regimen, with two exceptions:
  * mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
  * the pre-transplant dose of MPA will be half the standard post-transplant dose due to increased drug bioavailability in recipients with low glomerular filtration rate (GFR).
  Participants will be maintained on triple IS therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.
  Other Names: Regulatory Donor-Derived Dendritic Cells (DCreg)
  Arms: DCreg:2.5 to 5.0 million cells/kg+SOC

SUMMARY:
This study will evaluate the safety and feasibility of treatment involving a single infusion of donor-derived regulatory dendritic cells (DCreg) in first time, living donor renal transplant recipients.

DCreg will be prepared from monocytes obtained by leukapheresis from prospective (non-mobilized) living kidney donors and infused into the respective recipients 7 days before renal transplantation. This study will enroll 28 subjects (14 recipients, 14 donors). The duration of follow-up will be:

* 1 week following the leukapheresis procedure for donors and
* 2 years following their DCreg infusion for kidney recipients.

DETAILED DESCRIPTION:
This clinical trial is a single-center, open-label, dose-escalation, phase 1 study, enrolling N=14 de novo kidney transplant recipients and their respective living donors. The study objective is to evaluate the safety and feasibility of a single infusion of donor-derived regulatory dendritic cell (DCreg) treatment.

Transplant recipients will receive combination immunosuppressive agents according to the site's Standard of Care (SOC) regimen, with two exceptions:

* mycophenolic acid (MPA) will be initiated 7 days before transplant, at the time of donor DCreg infusion, instead of on the day of transplant; and
* the pre-transplant dose of MPA will be half the standard post-transplant dose, due to increased drug bioavailability in recipients with low kidney function defined by glomerular filtration rate (GFR).

Consequently, participants will be maintained on triple immunosuppressive therapy with MPA, tacrolimus, and prednisone after transplant, a combination regimen widely applied as SOC at many transplant centers in North America and worldwide.

Note: Participants will not be withdrawn from known effective therapy for the purpose of participating in this research.

ELIGIBILITY:
Inclusion Criteria:

Donor Eligibility Criteria:

* Able to understand and provide informed consent;
* Male or female >/= 18 years of age
* Meets all standard institutional criteria for kidney donation and Health Agency criteria for kidney donation;
* For females of childbearing potential, a negative urine or serum pregnancy test;
* Negative for Human Immunodeficiency Virus type 1 (HIV) -1 (antigen and Nucleic Acid Testing (NAT)), HIV-2, Human T-cell leukemia virus type 1 (HTLV-1), and HTLV-2;
* Negative for hepatitis C (antibody and NAT), hepatitis B (surface antigen and core antibody), and Treponema pallidum infection;
* Negative for West Nile Virus;
* Negative health history for Creutzfeldt-Jakob disease;
* No live vaccines within 8 weeks prior to leukapheresis;
* No medical condition(s) that the investigator deems incompatible with participation in the trial; and
* No use of investigational drugs within 12 weeks of participation.

Recipient Inclusion Criteria:

* Must be able to understand and provide informed consent;
* Is >/= 18 years old at the time of informed consent;
* Is undergoing a living donor renal transplant;
* For females of childbearing potential, a negative urine or serum pregnancy test upon study entry
* The candidate agrees to use contraception with a method that is more than 80% effective (see FDA Office of Women's Health (http://www.fda.gov/birthcontrol). Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) to be used from one month before study treatment begins until one month after study completion;
* Cytomegalovirus (CMV) seropositive or, if CMV seronegative must be receiving a kidney from a CMV seronegative donor;
* Has a negative purified protein derivative (PPD) or negative testing for tuberculosis using an approved IGRA blood test, such as QuantiFERON®-Gold TB or T-SPOT-TB assay OR has completed treatment for latent tuberculosis and has a negative chest x-ray. PPD or IGRA testing must occur within 52 weeks before transplant. These requirements apply as well to prior recipients of Bacille Calmette-Guérin (BCG) vaccination;
* Meets all standard institutional and Health Agency criteria for kidney transplant.
* Vaccines up to date as per DAIT guidance for patients in transplant trials (Refer to Manual of Operations).

Study Exclusion Criteria:

* Panel Reactive Antibody (PRA >20%);
* Positive T or B Cell Flow Crossmatch prior to transplant;
* Presence of donor specific antibody (DSA) ≥ to mean fluorescence intensity (MFI) of 1000, or DSA between 500 and 1000, if a specific shared epitope pattern is present;
* Recipient of multi-organ transplant;
* Any prior renal or extra-renal transplant with HLA class II antigen mismatch shared with prior organ;
* Epstein-Barr Virus (EBV) Immunoglobulin G (IgG) negative if the donor is EBV positive;
* Seropositivity for HIV-1, hepatitis B core antigen, or hepatitis C virus (HCV) antibody (if hepatitis C antibody positive, confirm negative infection by HCV RNA), or positivity for hepatitis B surface antigen;
* History of malignancy witin the past 5 years unless standard institutional criteria detailed in Appendix 6 have been met;
* High risk for recurrence of renal disease: Hemolytic Uremic Syndrome Thrombotic Thrombocytopenic Purpura (HUS-TTP); Focal Segmental Glomerular Sclerosis (FSGS); or Aggressive native kidney disease.
* Compensated and decompensated cirrhosis of liver and/or portal hypertension;
* Chronic Obstructive Pulmonary Disease requiring nasal oxygen, and/or pulmonary hypertension (mean pulmonary pressure >45mm/hg);
* Any history of stroke with neurological deficit;
* Any condition that, in the opinion of the investigator, confers excessive risk for participation in this phase 1 study;
* Presence of a condition that requires treatment with an immunosuppressive agent, other than a physiologic dose of corticosteroid;
* Live vaccines within 8 weeks prior to transplant;
* Use of investigational drugs within 12 weeks of participation;
* Woman receiving a kidney from a man who has fathered her child(ren), whether or not carried to term; or
* Woman receiving a kidney from her biological child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome: Proportion of Participants who Experience any of the Pre-Specified Safety Events | Seven Days Prior to Transplant Surgery(e.g. Day of Regulatory Dendritic Cells (DCreg) Infusion) up to 1-Year Post-Transplant
  Safety will be assessed by summarizing the proportion of participants who experience any of the following events from the initiation of the regulatory dendritic cells (DCreg) infusion administered 7 days prior to kidney transplant to 1 year post-transplant:
  * Recipient death attributed to receipt of DCreg,
  * NCI-CTCAE Grade 4 or higher DCreg infusion reaction,
  * NCI-CTCAE Grade 4 or higher infection,
  * Malignancy other than non-melanoma skin cancer,
  * Pre-transplant Donor Specific Antibodies (DSA),
  * Post-transplant DSA,
  * Biopsy-proven acute rejection (BPAR) by BANFF 2017 criteria (grade ≥2A), or
  * Non-surgical graft loss.
    * Reference: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0).

SECONDARY OUTCOMES:
Incidence of Death Attributed to Participant Receipt of Regulatory Dendritic Cells (DCreg) | Seven Days Prior to Transplant Surgery (e.g. Day of Regulatory Dendritic Cells (DCreg) Infusion) up to 1-Year Post-Transplant
  The occurrence of death among participants who receive DCreg treatment.
Incidence of Adverse Event: CTCAE Grade 4 or Higher Infusion Reaction | Seven Days Prior to Transplant Surgery (e.g. Day of Regulatory Dendritic Cells (DCreg) Infusion) up to 1-Year Post-Transplant
  The number of Grade 4 or higher infusion reaction(s) among participants who receive regulatory dendritic cells (DCreg) infusion, graded in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0).
Incidence of Adverse Event:CTCAE Grade 4 or Higher Infection | Seven Days Prior to Transplant Surgery (e.g. Day of Regulatory Dendritic Cells (DCreg) Infusion) up to 1-Year Post-Transplant
  The number of Grade 4 or higher infection(s) among participants who receive regulatory dendritic cells (DCreg) infusion, graded in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0).
Incidence of Adverse Event: Malignancy | Seven Days Prior to Transplant Surgery(e.g. Day of Regulatory Dendritic Cells (DCreg) Infusion) up to 1-Year Post-Transplant
  The number of malignancies among participants who receive regulatory dendritic cells (DCreg) infusion. Not included in this incidence outcome: non-melanoma skin cancer(s).
Incidence of Pre-Transplant Donor Specific Antibodies (DSA) | Baseline (Seven Days Prior to Transplant Surgery, "Pre" -Regulatory Dendritic Cells (DCreg)) Infusion) up to within 48 Hours of Transplant
  The number of pre-transplant DSA among participants occurring after DCreg infusion and before transplant.
Incidence of Post-Transplant Donor Specific Antibodies (DSA) | Day 0 (Transplant Surgery) up to 1-Year Post-Transplant
  A de novo DSA occurring within the first year post-transplant.
Incidence of Biopsy-Proven Acute Rejection | Day 0 (Transplant Surgery) up to 1-Year Post-Transplant
  Acute kidney allograft rejection is defined by a kidney (renal) allograft biopsy classification of grade 2A or higher. Classification method: Banff 2013. The Banff 2013 classification for antibody-mediated rejection is a recognized standard in renal allograft pathology.
Incidence of Non-Surgical Graft Loss | Day 0 (Transplant Surgery) up to 1-Year Post-Transplant
  Graft loss not associated with the transplant surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amit D. Tevar, MD, FACS, Study Chair — University of Pittsburgh: Starzl Transplantation Institute
Locations (1):
- University of Pittsburgh, Starzl Transplantation Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190
- [Background] Haas M. The Revised (2013) Banff Classification for Antibody-Mediated Rejection of Renal Allografts: Update, Difficulties, and Future Considerations. Am J Transplant. 2016 May;16(5):1352-7. doi: 10.1111/ajt.13661. Epub 2016 Feb 4. PMID 26696524
- See also: NIH NCI Common Terminology Criteria for Adverse Events (CTCAE) — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm